CLINICAL TRIAL: NCT06796010
Title: Assessment of the Protective Effect of Four Sunscreens on Visible Light Induced Pigmentation Compared with an Untreated Control Zone
Brief Title: Photoprotection Efficacy of Four Sunscreen Formulas Under Visible Light Exposure
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-07408 / CPC-3571
Record Dates: First submitted 2025-01-14; First posted 2025-01-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Visible Light Exposure; Healthy Back Skin
Keywords: Photoprotection; Sunscreen; Visible Light (VL); Pigmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Product 1: The test product 1 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 2: The test product 2 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 3: The test product " was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 4: The test product 4 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Untreated zone: non-treated control zone
  Interventions: Other: Visible Light Exposure - Untreated zone

INTERVENTIONS:
Other: Visible Light Exposure - Treated zones — The treated zones were exposed to Visible Light to induce skin pigmentation (144J/cm2), 15 to 30 minutes after application.
  Groups: Product 1; Product 2; Product 3; Product 4
Other: Visible Light Exposure - Untreated zone — The untreated zone was exposed to Visible Light to induce skin pigmentation (144J/cm2), as the same time as the treated zones.
  Groups: Untreated zone

SUMMARY:
To evaluate the protective effect of four sunscreens on the pigmentation caused by visible light in comparison to an untreated control zone in healthy volunteers.

DETAILED DESCRIPTION:
The sunscreens usually used as photoprotectors are known to protect in the UV domain (UVB and UVA). However, until recently visible light (400-700 nm) was considered as devoid of any photobiological effects on cutaneous tissue. Over the last two decades, with the development of photodynamic therapies and various dermatological treatments using visible laser light, several studies have reconsidered the cutaneous effect of visible light on the skin, in particular the induction of pigmentation.

The aim of this study was to assess the ability of sunscreens with a protective efficacy in the UV domain to prevent the pigmentation induced by Visible Light.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects of both sexes aged 18 - 50 years old, having a phototype IIIb, IV or V according to Fitzpatrick classification,
2. Subject with an ITA° (Individual Typologic Angle calculated value) between -20° and 28° at the screening visit,
3. Healthy subjects based on physical examination and compatibility of medical history with the study content,
4. Women of childbearing potential using adequate contraception (oral contraception, intra-uterine devices, contraceptive implants or vaginal rings, tubal sections or ligations, condoms) for at least 1 month prior to first visit and agree to continue adequate contraception during the entire duration of the study,
5. Women of non-childbearing potential (menopausal with one year without bleeding, hysterectomy, bilateral ovariectomy),
6. Subjects having signed a written informed consent form and dated before any study procedure begins.
7. Subjects should be willing to actively cooperate during the study duration and willing to complete the study,
8. Subject affiliated to the social security system (in accordance with the French Law 2004-806 and its implementing decree n°2006-477 of 26 April 2006).

Exclusion Criteria:

1. Female who is pregnant or breast feeding or planning a pregnancy during the study,
2. Subject having an underlying known disease, or surgical, physical, or medical condition that, in the opinion of the Investigator might interfere with the interpretation of the clinical trial results such as:

   1. History of recurrent dermatologic conditions (e.g., psoriasis, eczema, urticaria…) or suspicion/history of allergy to cosmetics,
   2. Any systemic or local disease pathology
   3. Skin abnormality (scars, excessive hair, tattoos…) at the level of the test zones (middle part of the back),
3. Subject who has been overexposed to natural (sun) or artificial ultraviolet (tanning lamps) in the last month prior the first visit or who plans a such exposure during the study;
4. Subject having history or presenting pathologies induced or aggravated by sun exposure or having abnormal reactions to the sun (ex : photosensitive dermatitis, polymorphic light eruption, solar urticaria, systemic erythematous lupus, dermatomyositis),
5. Subject having taken a systemic treatment more than 5 days in the month preceding the inclusion (steroids, nonsteroidal anti-inflammatory drugs such as aspirin, antihistamine, insulin, hypertensors, antibiotics such as quinolones, tetracyclins, thiazids, fluoroquinolons and and photosensitizing treatment) or any treatment able to induce abnormal response to UV or visible light (vitamin A derivatives, psoralen, aminolevulinic acid etc.) or having plane to take these treatments during the study,
6. Subjects having applied a local treatment on the back for more than 2 days during the 2 weeks preceding inclusion (steroids, non-steroidal anti-inflammatories, antihistamines, antibiotics) and all other cosmetic products in the previous 24 hours,
7. Subject having antecedents of clinically significant allergy, particularly to study product components,
8. Subjects requiring enhanced protection (deprived of liberty, minors, under guardianship),
9. Subject being in a situation which, according to the Investigator, could interfere with an optimal participation in the study,
10. Subject currently participating or having participated in another clinical trial during the month preceding inclusion,
11. Subject under care of guardian or legal guardianship or subject hospitalized in a medical or social establishment for any reason,
12. Subject unable to communicate efficiently with the Investigator or being unable to follow the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers from 18 to 50 years old with phototype III to V according to the Fitzpatrick scale and with an ITA° between -28° to 20° at Screening
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2019-11-23 (Actual)

PRIMARY OUTCOMES:
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4, Day 5 (24 hours after each Visible Light exposure) and Day 12
  Individual Typologic Angle (ITA° - calculated value), • Pigmentation (Delta E, Delta L* and Delta b* - calculated values), • Erythema (Delta a* - calculated value).

SECONDARY OUTCOMES:
Clinical investigator's assessment by using clinical scale | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4, Day 5 (24 hours after each Visible Light exposure) and at Day 12..
  Visual scoring of pigmentation, using a pigmentation 11-point scale with 0 (No pigmentation), 1 (Doubtful), 2 (Very pale brown -), 3 (Very pale brown), 4 (Very pale brown +), 5 (Pale brown -), 6 (Pale brown), 7 (Pale brown +), 8 (Brown -), 9 (Brown), 10 (Brown +) Visual scoring of erythema, using an erythema 4-point scale with 0 (Absent), 0.5 (Doubtful), 1 (Weak but well-defined erythema), 2 (Moderate), 3 (Severe)
Safety / Local Tolerance | From the informed consent signature date until the end of the study (Day 12).
  Safety was assessed by recording Adverse Events, including cutaneous reactions (local intolerance) assessed using the following 5-point score system:
  0 (no sign/symptom of local intolerance); 0.5 (doubtful sign/symptom of local intolerance); 1 (mild sign/symptom of local intolerance); 2 (moderate sign/symptom of local intolerance); 3 (severe sign/symptom of local intolerance)

CONTACTS AND LOCATIONS:
Locations (1):
- CPCAD (Centre de Pharmacologie Clinique Appliquée à la Dermatologie), Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renoux P, Jouni H, Laloux C, Touti R, Vieu DL, Lamarche F, Santos SM, Bernerd F, Marionnet C. Visible Light-Induced Pigmentation: Improved In Vivo Methodology for Measuring Efficacy of 30 Products in 9 Randomised Controlled Trials and Correlation With In Vitro Assessment. Exp Dermatol. 2025 Sep;34(9):e70167. doi: 10.1111/exd.70167. PMID 40922539